CLINICAL TRIAL: NCT05466279
Title: Department of Anesthesiology, Cancer Hospital of the University of Chinese Academy of Sciences（Zhejiang Cancer Hospital), Research Center for Neuro-Oncology Interaction , Institute of Basic Medicine and Cancer, Chinese Academy of Sciences.
Brief Title: The Role of Remazolam in Reducing the Incidence of Postoperative Delirium in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fang Jun (Other)
Responsible Party: Sponsor-Investigator, Fang Jun, Clinical Professor, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-2020-344
Record Dates: First submitted 2022-07-13; First posted 2022-07-20 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Propofol; Midazolam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remazolam general anesthesia group (R group) (Experimental)
  Interventions: Drug: remazolam
- Propofol + midazolam general anesthesia control group (group P) (Active Comparator)
  Interventions: Drug: Propofol; Drug: Midazolam

INTERVENTIONS:
Drug: remazolam — Remimazolam is a new drug innovation in anesthesia. It combines the properties of two unique drugs already established in anesthesia - Midazolam and remifentanil.
  Arms: Remazolam general anesthesia group (R group)
Drug: Propofol — Propofol (2,6-diisopropylphenol) is a hypnotic agent that is used as an induction agent and as a maintenance anaesthetic delivered by continuous i.v. infusion or intermittent i.v. bolus
  Arms: Propofol + midazolam general anesthesia control group (group P)
Drug: Midazolam — Midazolam, like diazepam, is a benzodiazepine anxiolytic drug, which is used to treat anxiety, but its t ½ is much shorter or only about 2 h compared with 43 h for diazepam
  Arms: Propofol + midazolam general anesthesia control group (group P)

SUMMARY:
This study is a prospective, randomized, controlled trial.The selected patients were randomly divided into remazolam general anesthesia group and propofol + midazolam general anesthesia control group according to computer randomization method. There were 65 patients in each group. Remazolam general anesthesia group (R group): Remazolam 0.4 mg/kg for rapid induction of loss of consciousness for anesthesia induction and 1 mg/kg/h for maintenance. Propofol + midazolam general anesthesia control group (group P): propofol 1.5 mg/kg + midazolam 0.05 mg/kg slow intravenous push until the patient's consciousness disappeared, then propofol 4-8 mg/kg/h Anesthesia was maintained. Except for different sedative drugs, the analgesic and muscle relaxant medication regimens were the same between the two groups. In the study, the application of inhaled anesthetics, other benzodiazepines and anticholinergic drugs was restricted, and the mean arterial pressure during the operation was kept above 60 mmHg to avoid perioperative hypotension, hypoxemia, and hypercapnia. Warm measures were used to maintain the patient's intraoperative body temperature above 36.0 °C. POD assessment was performed on the day before surgery and on days 1-7 after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with limited abdominal tumor surgery (age ≥65 years)
* ASA classification I-III.

Exclusion Criteria:

* Refusing to participate in the study
* Patients with severe arrhythmia or cardiac dysfunction (EF<35%)
* A clear history of neurological and psychiatric disorders before surgery or long-term use of sedatives or antidepressants
* History of alcoholism or drug dependence
* History of brain surgery or trauma
* Severe vision or hearing impairment
* Inability to cooperate with the completion of cognitive function tests

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 131 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Postoperative, 7 days
  Proportion of patients with postoperative delirium among enrolled patients. The incidence of delirium during recovery was assessed by the Confusion Assessment Method-ICU (CAM-ICU). The assessment time points were: 10 minutes, 30 minutes after entering the anesthesia recovery room (or exiting the recovery room).
  The incidence of delirium within 7 days after surgery was assessed using 3D-CAM to assess whether patients had delirium.

SECONDARY OUTCOMES:
Intraoperative awareness rate | Postoperative, 24 hours
  The modified Brice interview over quality assurance techniques in detecting intraoperative awareness with explicit recall.
Intraoperative hemodynamic stability | Intraoperative, 6 hours
  The change curve of intraoperative mean arterial blood pressure and heart rate
Richard-campbell Sleep Questionnaire Score | Postoperative, 3 days
  Richards-Campbell Sleep Questionnaire (RCSQ) is a five-item、 visual analogue scale was designed for assessing sleep quality of patients
Perioperative nutritional status score table(PONS) | Baseline, 1 year
  Perioperative Nutrition Screen (PONS). This algorithmic approach is used to identify perioperative malnutrition risk and guide perioperative nutrition intervention. BMI, body mass index
Modified frailty rating scale | Baseline, 1 year
  Modified Frailty Index Frailty index is an important predictive variable in emergency general surgery patients older than 60 years. The modified frailty index can be used to evaluate risk of both morbidity and mortality in these patients.
Postoperative hospital stay | Postoperative, 3 months
  Taking the operation day as the starting point, calculating the length of stay in the hospital after the operation
Postoperative nausea and vomiting | Postoperative, 7 days
  The proportion of patients with nausea and vomiting within 7 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hanzhou, China

IPD SHARING:
Plan to Share IPD: No